CLINICAL TRIAL: NCT03239444
Title: Visualization of Human Cardiovascular Anatomy With Foresight Intracardiac Echocardiography (ICE) System
Brief Title: Foresight Intracardiac Echocardiography System (ICE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Conavi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: EXT-001-1.5
Record Dates: First submitted 2017-07-24; First posted 2017-08-04 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2017-07

CONDITIONS: Atrial Fibrillation
Keywords: ICE; Ablation; Trans-septal; Septum; Echocardiography
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Assigned Intervention (Other): Device: Foresight ICE System The Foresight ICE System is composed of a sterile, single-use catheter intended to operate with a Foresight ICE PIM and Hummingbird console. The Foresight ICE system will be used in guiding the physician during the trans-septal puncture and provide physiological information during the course of the procedure.
  Interventions: Device: Intracardiac echocardiography imaging

INTERVENTIONS:
Device: Intracardiac echocardiography imaging — Wide visualization of the the heart anatomy and additional devices used during atrial fibrillation ablation procedures.

SUMMARY:
This study will evaluate the efficacy of the Foresight Intracardiac Echocardiography system ,with improved image quality, in guiding trans-septal punctures during atrial fibrillation ablation procedures.

DETAILED DESCRIPTION:
The study will recruit 10 patients at a single center.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years old.
* Patient is undergoing an atrial fibrillation ablation procedure.
* Patient has a transesophageal echocardiogram (TEE) within the 48 hours prior to ablation procedure to rule out left atrial thrombus.
* Patient provides informed, written consent for participation in the study.

Exclusion Criteria:

* Patients in whom placement of an ICE catheter in the right atrium for adequate atrial visualization is not technically feasible (as evaluated and determined by the physician/study investigator performing the procedure).
* Patients in whom transseptal puncture is relatively contraindicated.
* Patients in whom left atrial clot or dense spontaneous contrast is identified on TEE, which would increase thromboembolic risk.
* Women of child bearing potential, in whom pregnancy cannot be excluded.
* Patients unable to grant informed, written consent for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2018-12-24 (Actual); Study Completion 2018-12-24 (Actual)

PRIMARY OUTCOMES:
Evaluation of the study device for guiding transseptal puncture in order to gain access to the left atrium of the heart during an ablation procedure in patients suffering with atrial fibrillation. | For each patient, the individual physician satisfaction survey will be completed on the day of the procedure.
  The ability of the study device to identify the atrial septum during transseptal puncture will be evaluated by the physician on the day of the procedure and captured in the individual case report form. This will be based on the objective finding of whether the transseptal puncture was performed (Yes or No) under study device guidance. This information will be gathered for each patient in the individual case report form and presented qualitatively and as quantitative measures (percentage success).

SECONDARY OUTCOMES:
Collection of first human images with Conavi's Foresight System. | An individual physician satisfaction survey will be completed for each case on the day of the procedure.
  The Conavi's Foresight System will be utilized to capture images of relevant human cardiac anatomical landmarks (e.g. crista terminalis, tricuspid valve, coronary sinus) while the catheter will be manipulated inside the heart during the procedure. The physician satisfaction survey will ask the physician to specifically tabulate structures that could be identified in a binary yes/no format.
  This kind of information will be gathered for each patient in the individual physician satisfaction surveys and presented qualitatively.

CONTACTS AND LOCATIONS:
Overall Officials: Atul Verma, MD, Principal Investigator — Southlake Regional Health Center, Newmarket, Ontario, Canada, L3Y2P6
Locations (1):
- Southlake Regional Health Centre, Newmarket, Ontario, Canada